CLINICAL TRIAL: NCT00745121
Title: An Open, Prospective, Non-randomized, Controlled, Multicenter Study to Evaluate Clinical Outcome of the ASTRA TECH Implant System, OsseoSpeed™ Implant in Women Over 60 Years of Age With Osteoporosis/Osteopenia
Brief Title: Study Evaluating ASTRA TECH Implant System, OsseoSpeed™ Implants in the Upper Jaw in Women With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-OSS-0007
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Postmenopausal Osteoporosis; Osteopenia; Jaw, Edentulous, Partially
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-A, Osteoporosis/osteopenia (Experimental): Patients with osteoporosis/osteopenia.
  Interventions: Device: OsseoSpeed™
- Group-B, Control (Experimental): Control (non-osteoporotic/-osteopenic patients).
  Interventions: Device: OsseoSpeed™

INTERVENTIONS:
Device: OsseoSpeed™ — ASTRA TECH Implant System, OsseoSpeed™ implants Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm

SUMMARY:
The overall objective of the study is to compare treatment with the ASTRA TECH Implant System, OsseoSpeed™ implant in the maxilla of postmenopausal women with and without systemic osteoporosis. The hypothesis is that there will be no difference in marginal bone level alterations between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Postmenopausal women aged 60 years and over
* In need of 2-8 implants in maxilla
* A history of edentulism in the area of implant treatment of at least 6 months.
* A Bone Mineral Density (BMD) value suitable either for group A or group B:
* Group A (Osteoporosis/osteopenia): BMD at least 2 standard deviations (SD) below mean peak bone density of young adults for the spine and total hip (T-score = -2 SD or less). Absolute values (g/cm2) will be used.
* Group B (Control): BMD not more than 1 standard deviation below mean peak bone density of young adults for the spine and total hip (T-score = -1 SD or more). Absolute values (g/cm2) will be used.

Exclusion Criteria:

* Unlikely to be able to comply with study procedures, as judged by the investigator.
* Untreated, uncontrolled caries and/or periodontal disease
* Known or suspected current malignancy
* History of chemotherapy within 5 years prior to surgery
* History of radiation in the head and neck region
* History of other metabolic bone diseases, e.g. Paget's disease, hyperparathyroidism, fibrous dysplasia or osteomalacia
* A medical history that makes implant insertion unfavourable
* Need for systemic corticosteroids
* Current or previous use of intravenous bisphosphonates (esp. zoledronic acid)
* Current or previous use of oral bisphosphonates
* History of bone grafting and/or sinus lift in the planned implant area
* Current need for bone grafting and/or sinus lift in the planned implant area
* Present alcohol and/or drug abuse
* Involvement in the planning and conduct of the study (applies to both Astra Tech AB staff or staff at the study site)
* Previous enrolment in the present study.
* Participation in a clinical study during the last 6 months.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-07-16; Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quirynen, Prof., Dr., Principal Investigator — KU Leuven
Locations (4):
- Department of Periodontology, Faculty of Medicine, Catholic University of Leuven, Leuven, Belgium
- Zahnklinik, Würzburg, Germany
- Sweden (2):
  - Department of Oral and Maxillofacial Surgery, Gothenburg University, Gothenburg
  - Käkkirurgiska kliniken, Akademiska sjukhuset, Uppsala

REFERENCES:
- [Result] Merheb J, Temmerman A, Coucke W, Rasmusson L, Kubler A, Thor A, Quirynen M. Relation between Spongy Bone Density in the Maxilla and Skeletal Bone Density. Clin Implant Dent Relat Res. 2015 Dec;17(6):1180-7. doi: 10.1111/cid.12228. Epub 2014 Jun 6. PMID 24909074
- [Result] Merheb J, Temmerman A, Rasmusson L, Kubler A, Thor A, Quirynen M. Influence of Skeletal and Local Bone Density on Dental Implant Stability in Patients with Osteoporosis. Clin Implant Dent Relat Res. 2016 Apr;18(2):253-60. doi: 10.1111/cid.12290. Epub 2016 Feb 10. PMID 26864614
- [Result] Temmerman A, Rasmusson L, Kubler A, Thor A, Quirynen M. An open, prospective, non-randomized, controlled, multicentre study to evaluate the clinical outcome of implant treatment in women over 60 years of age with osteoporosis/osteopenia: 1-year results. Clin Oral Implants Res. 2017 Jan;28(1):95-102. doi: 10.1111/clr.12766. Epub 2016 Jan 7. PMID 26744141
- [Result] Temmerman A, Rasmusson L, Kubler A, Thor A, Merheb J, Quirynen M. A Prospective, Controlled, Multicenter Study to Evaluate the Clinical Outcome of Implant Treatment in Women with Osteoporosis/Osteopenia: 5-Year Results. J Dent Res. 2019 Jan;98(1):84-90. doi: 10.1177/0022034518798804. Epub 2018 Sep 11. PMID 30205020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 103 participants were enrolled in the study (provided written informed consent).
Pre-assignment Details: 55 of the enrolled participants became screening failures and were excluded from the study before implant installation.
  The baseline population consist of all participants that had at least one implant installed, a total of 48 participants.
Units Other Than Participants: Implants
Groups:
- Group-A, Osteoporosis/Osteopenia: Patients with osteoporosis/osteopenia.
  Receiving OsseoSpeed™: ASTRA TECH Implant System, OsseoSpeed™ implants Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm
- Group-B, Control: Control (non-osteoporotic/-osteopenic patients).
  Receiving OsseoSpeed™: ASTRA TECH Implant System, OsseoSpeed™ implants Ø 3.5, 4, 4.5, 5.0 mm in lengths of 8, 9, 11, 13, 15, 17 and 19 mm
Period: Overall Study
Arm/Group | Group-A, Osteoporosis/Osteopenia | Group-B, Control
Started | 20; 63 Implants | 28; 85 Implants
Completed | 11; 37 Implants | 26; 77 Implants
Not Completed | 9; 26 Implants | 2; 8 Implants
Not completed — Death | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Population: A total of 103 participants were enrolled in the study (provided written informed consent).
  55 of those participants became screening failures and were excluded from the study before implant installation.
  The baseline population consist of all participants that had at least one implant installed, a total of 48 participants.
Units Other Than Participants: Implants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-A, Osteoporosis/Osteopenia | Group-B, Control | Total
Number analyzed (Participants) | 20 | 28 | 48
Number analyzed (Implants) | 63 | 85 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (6.18) | 64.9 (4.10) | 66.8 (5.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 19 | 28 | 47
  South American Indian (Chile) | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Sweden | 10 | 9 | 19
  Belgium | 5 | 13 | 18
  Germany | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Level Alterations
Description: Marginal Bone Level determined from radiographs and expressed as the difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal Bone Level expressed in millimeters at the 5 year follow-up visit compared to values obtained at time of loading of the permanent restoration (baseline).
Time Frame: Evaluated at time of loading of the permanent restoration and at the 5 years follow-up after loading.
Population: In group A, 11 subjects (38 implants) completed the 5-year follow-up visit. In group B, 26 subjects (79 implants) completed the 5-year follow-up visit.
  Three radiographs were not possible to evaluate, giving an overall number of 37 subjects (114 implants) as basis for the analysis of Marginal Bone Level Change.
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: Implants
Arm/Group | Group-A, Osteoporosis/Osteopenia | Group-B, Control
Number analyzed (Participants) | 11 | 26
Number analyzed (Implants) | 37 | 77
millimeter | -0.15 (0.50) | -0.06 (0.89)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Group-A, Osteoporosis/Osteopenia | Group-B, Control
All-Cause Mortality (participants affected / at risk) | 3/20 | 0/28
Serious Adverse Events (participants affected / at risk) | 6/20 | 5/28
Other Adverse Events (participants affected / at risk) | 2/20 | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-A, Osteoporosis/Osteopenia (N=20) | Group-B, Control (N=28)
Death, reason unknown (General disorders) | 3 (3) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Pancreatic cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cerebral colloid cyst (Nervous system disorders) | 0 (0) | 1 (1)
Removal of gall bladder (gallstone related) (Hepatobiliary disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Knee injury (due to a fall) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Operation (artificial shoulder joint) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Breast surgery (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-A, Osteoporosis/Osteopenia (N=20) | Group-B, Control (N=28)
Dental bridge loose (Product Issues) | 2 (2) | 0 (0) — the dental bridge screws connecting the implant abutment to the restoration coming loose
Fracture connecting bar (Product Issues) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-01-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT00745121/Prot_SAP_000.pdf